CLINICAL TRIAL: NCT04770376
Title: Prospective Pilot Study for the Evaluation of the Predictive Value of Blood Levels of Angiopoietin 1 (ANG1) and Endothelial Internal Tunica Cell Kinase 2 (TiE2) in Patients With Ovarian Cancer Treated With Chemotherapy Associated to bevAcizumab
Brief Title: Evaluation of the Predictive Value of Blood Levels of Angiopoietin 1 and Endothelial Internal Tunica Cell Kinase 2 in Patients With Ovarian Cancer Treated With Chemotherapy Associated to Bevacizumab
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Ospedale SS Giovanni e Paolo, Venezia (Unknown)
Responsible Party: Principal Investigator, Claudio Zamagni MD, MD Medical Oncologist, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: PANGEA
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; angiopoietin 1; tunica interna endothelial cell kinase 2; VEGF; bevacizumab
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: patients treated with chemotherapy (I-II line) associated to bevacizumab: Quantification of biomarkers will be performed on 100 patients treated with bevacizumab through the collection of the following samples at different timepoints: 1 serum sample; 2 CTAD plasma samples; 2 K2EDTA plasma samples. The samples will be collected as follows: before the start of chemotherapy; 3 weeks after start of chemotherapy, before start of treatment with bevacizumab; 9 weeks after start of chemotherapy; 15 weeks after start of chemotherapy; 52 weeks after start of chemotherapy; at progression of disease.
  Interventions: Other: Observational study. Blood samples will be collected at scheduled blood draws performed as per clinical practice before each cycle of chemotherapy.
- Cohort B: patients treated with chemotherapy (I-II line, not associated to antiangiogenic drugs): Quantification of biomarkers will be performed on 50 patients treated with chemotherapy through the collection of the following samples at different timepoints: 1 serum sample; 2 CTAD plasma samples; 2 K2EDTA plasma samples. The samples will be collected as follows: before the start of chemotherapy; 3 weeks after start of chemotherapy, before start of treatment with bevacizumab; 9 weeks after start of chemotherapy; 15 weeks after start of chemotherapy; 52 weeks after start of chemotherapy; at progression of disease.
  Interventions: Other: Observational study. Blood samples will be collected at scheduled blood draws performed as per clinical practice before each cycle of chemotherapy.

INTERVENTIONS:
Other: Observational study. Blood samples will be collected at scheduled blood draws performed as per clinical practice before each cycle of chemotherapy. — Collection of blood samples during blood draws performed before each cycle of chemotherapy as per clinical practice.

SUMMARY:
This is a monocentric prospective observational pilot study of translational research in women with advanced ovarian epithelial cancer. The main purpose of this study is to evaluate the predictive value of response to treatment with bevacizumab of the circulating levels of Ang1, Tie2 and VEGF before start of therapy. Secondary aims of the study are to explore the predictive value of response / resistance to bevacizumab of changes in circulating levels of Ang1 and Tie2 during treatment and at progression of disease, and to explore the possible role of circulating VEGF in the modulation of bioavailability of bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Diagnosis of histologically confirmed advanced epithelial ovarian carcinoma
* Women eligible for treatment with a chemotherapy regimen in combination to bevacizumab (Cohort A)
* Women eligible for treatment with a chemotherapy regimen not associated to antiangiogenic drugs (Cohort B)
* Evaluable disease according to RECIST 1.1 criteria
* Patient informed consent signature prior to any study-specific procedure

Exclusion Criteria:

* History of other malignancy within 5 years prior to study entry (except for cutaneous basal cell carcinoma or adequately treated carcinoma in situ of the cervix ).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample size of 100 patients with advanced epithelial ovarian carcer is expected to be enrolled in Cohort A (I-II line of chemotherapy associated to bevacizumab) and 50 patients with advanced epithelial ovarian carcer is expected to be enrolled in Cohort B (I-II line of chemotherapy, not associated to antiangiogenic drugs)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
relationship between Ang1 and Tie2 values and response to treatment with bevacizumab | Before start of chemotherapy
  Relationship between baseline values of Ang1 and Tie2 (considered individually or combined with each other) and response to treatment with bevacizumab (according to RECIST 1.1 criteria).
relationship between VEGF values and response to treatment with bevacizumab | Before start of chemotherapy
  Relationship between baseline values of endogenous VEGF (plasma CTAD levels) and released by platelets during the clot phase (serum levels) and response to treatment with bevacizumab.

SECONDARY OUTCOMES:
relationship between Ang1 and Tie2 levels | from baseline (before start of chemotherapy) to 52 weeks from start of chemotherapy or progression of disease
  relationship between Ang1 and Tie2 levels at baseline, during chemotherapy administration and at progression of disease.
anticipation of diagnosis of progression of disease | from baseline (before start of chemotherapy) to 52 weeks from start of chemotherapy or progression of disease
  possible anticipation of diagnosis of progression of disease through evaluation of Ang1 and Tie2
VEGF evaluation | from baseline (before start of chemotherapy) to 52 weeks from start of chemotherapy or progression of disease
  Evaluation of free VEGF, bevacizumab-bound VEGF and available bevacizumab in relation to clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Zamagni, MD, Principal Investigator — Policlinico S.Orsola-Malpighi, SSD Oncologia Medica Addarii
Locations (1):
- Azienda Ospedaliero-Universitaria di Bologna, Policlinico S. Orsola-Malpighi, SSD Oncologia Medica Addarii, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gadducci A, Lanfredini N, Sergiampietri C. Antiangiogenic agents in gynecological cancer: State of art and perspectives of clinical research. Crit Rev Oncol Hematol. 2015 Oct;96(1):113-28. doi: 10.1016/j.critrevonc.2015.05.009. Epub 2015 Jun 16. PMID 26126494
- [Background] Oliver KE, McGuire WP. Ovarian cancer and antiangiogenic therapy: caveat emptor. J Clin Oncol. 2014 Oct 20;32(30):3353-6. doi: 10.1200/JCO.2014.57.4574. Epub 2014 Sep 15. No abstract available. PMID 25225422
- [Background] Backen A, Renehan AG, Clamp AR, Berzuini C, Zhou C, Oza A, Bannoo S, Scherer SJ, Banks RE, Dive C, Jayson GC. The combination of circulating Ang1 and Tie2 levels predicts progression-free survival advantage in bevacizumab-treated patients with ovarian cancer. Clin Cancer Res. 2014 Sep 1;20(17):4549-4558. doi: 10.1158/1078-0432.CCR-13-3248. Epub 2014 Jun 19. PMID 24947924
- [Background] Zhou C, Clamp A, Backen A, Berzuini C, Renehan A, Banks RE, Kaplan R, Scherer SJ, Kristensen GB, Pujade-Lauraine E, Dive C, Jayson GC. Systematic analysis of circulating soluble angiogenesis-associated proteins in ICON7 identifies Tie2 as a biomarker of vascular progression on bevacizumab. Br J Cancer. 2016 Jul 12;115(2):228-35. doi: 10.1038/bjc.2016.194. Epub 2016 Jun 28. PMID 27351218
- [Background] Jayson GC, Zhou C, Backen A, Horsley L, Marti-Marti K, Shaw D, Mescallado N, Clamp A, Saunders MP, Valle JW, Mullamitha S, Braun M, Hasan J, McEntee D, Simpson K, Little RA, Watson Y, Cheung S, Roberts C, Ashcroft L, Manoharan P, Scherer SJ, Del Puerto O, Jackson A, O'Connor JPB, Parker GJM, Dive C. Plasma Tie2 is a tumor vascular response biomarker for VEGF inhibitors in metastatic colorectal cancer. Nat Commun. 2018 Nov 7;9(1):4672. doi: 10.1038/s41467-018-07174-1. PMID 30405103
- [Background] Ciccolini J, Serdjebi C, Barbolosi D, Lacarelle B, Barlesi F. Ang1 and Tie2 are predictive biomarkers for bevacizumab-letter. Clin Cancer Res. 2015 Feb 15;21(4):934. doi: 10.1158/1078-0432.CCR-14-2832. No abstract available. PMID 25691775
- [Background] Loupakis F, Falcone A, Masi G, Fioravanti A, Kerbel RS, Del Tacca M, Bocci G. Vascular endothelial growth factor levels in immunodepleted plasma of cancer patients as a possible pharmacodynamic marker for bevacizumab activity. J Clin Oncol. 2007 May 1;25(13):1816-8. doi: 10.1200/JCO.2006.10.3051. No abstract available. PMID 17470880